CLINICAL TRIAL: NCT01226186
Title: Self Medication With Oral Morphine After Total Knee Arthroplasty. A Randomised Controlled Trial Comparing Self Medication With Standard Nurse Dispensing. Is There a Difference in Morphine Consumption, Pain, Patient Satisfaction or Safety?
Brief Title: Self Medication With Oral Morphine After Total Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Collaborators: Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/H0505/77
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Arthroplasty, Knee Replacement; Pain Control
Keywords: Knee replacement; Pain control; Self medication
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse dispensed oral morphine solution. (Active Comparator)
  Interventions: Behavioral: Nurse dispensed oral morphine.
- Self medicated oral morphine solution. (Active Comparator)
  Interventions: Behavioral: Patient self medication of oral morphine.

INTERVENTIONS:
Behavioral: Nurse dispensed oral morphine. — Nurse will dispense oral morphine on request from the patient.
  Arms: Nurse dispensed oral morphine solution.
Behavioral: Patient self medication of oral morphine. — Patients will self medicate their oral morphine pain control solution following surgery.
  Arms: Self medicated oral morphine solution.

SUMMARY:
The study aims to compare two post operative pain management strategy's, traditional nurse dispensed pain control versus patient self medication. The investigators aim to establish if patients who self medicate have differing pain levels than those who take nurse dispensed oral morphine.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring total knee replacement surgery willing to provide written, informed consent.

Exclusion Criteria:

* Unable to safely self medicate.

Allergy to morphine.

Unable to provide consent.

Contraindication to the standardised anaesthetic or standard postoperative care.

Not consenting to an element of the standardised anaesthetic.

Pre-operative use of strong opiates e.g. Oramorph, MST, Oxynorm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To establish if patients who self medicate with oral morphine have differing pain levels than those who take nurse dispensed oral morphine. | one year

SECONDARY OUTCOMES:
To identify if patients who self medicate with oral morphine take a significantly different amount of morphine compared with those who take nurse dispensed oral morphine. | one year
To compare whether patients who self medicate with oral morphine have a significantly altered level of side effects compared with those who take nurse dispensed oral morphine. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Linton, Doctor, Principal Investigator — Poole Hospital NHS Foundation Trust
Locations (1):
- Derwent Unit, Royal Bournemouth Hospital., Bournemouth, Dorset., United Kingdom